CLINICAL TRIAL: NCT05811533
Title: Comparison of Spencer's Muscle Energy Technique and Post-facilitation Stretch in Patients With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/MS-PT/01496 Neelam
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Frozen Shoulder
Keywords: spencer Muscle energy technique; post facilitation; pain; range of motion
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spencer's MET with conventional therapy (Experimental): Patients will be asked to lie in a side lying position with the affected shoulder above. The therapist will stabilize the shoulder girdle with the proximal hand and the distal hand provided force into the restrictive barrier of shoulder in 7 different movements. During all the movements, patients will ask to use their muscle energy 20% against the slight resistance offered by the therapist for 3-5 seconds. The patient then asks to relax and exhale after that shoulder joint will move beyond the barrier to achieve the next barrier. After 20 sec of rest, this technique will be repeated 3-5 times
  Interventions: Other: Spencer's MET with conventional therapy
- Post-Facilitation Stretch with conventional therapy (Experimental): Muscle Energy Technique [Post Facilitation Stretch)] for the shoulder joint will be applied with 3 repetitions per set, 1 session per day. Patient will be instructed to perform a full strength contraction of the muscle to be stretch for 10 seconds. The muscle is then allow to fully relax, whereupon a rapid stretch of the affected muscle will be performed and will held in position by the physician for 15 sec. Patient will be asked to relax and whole cycle will be repeated.
  Interventions: Other: Post-Facilitation Stretch with conventional therapy

INTERVENTIONS:
Other: Spencer's MET with conventional therapy — Patients will be asked to lie in a side lying position with the affected shoulder above. The therapist will stabilize the shoulder girdle with the proximal hand and the distal hand provided force into the restrictive barrier of shoulder in 7 different movements. During all the movements, patients will ask to use their muscle energy 20% against the slight resistance offered by the therapist for 3-5 seconds. The patient then asks to relax and exhale after that shoulder joint will move beyond the barrier to achieve the next barrier. After 20 sec of rest, this technique will be repeated 3-5 times
  Arms: Spencer's MET with conventional therapy
Other: Post-Facilitation Stretch with conventional therapy — Muscle Energy Technique [Post Facilitation Stretch)] for the shoulder joint will be applied with 3 repetitions per set, 1 session per day. Patient will be instructed to perform a full strength contraction of the muscle to be stretch for 10 seconds. The muscle is then allow to fully relax, whereupon a rapid stretch of the affected muscle will be performed and will held in position by the physician for 15 sec. Patient will be asked to relax and whole cycle will be repeated
  Arms: Post-Facilitation Stretch with conventional therapy

SUMMARY:
Adhesive capsulitis is one of the most common problems of the upper limb. Adhesive capsulitis (AC) and frozen shoulder syndrome (FSS) are two terms that have been used to describe a painful and stiff shoulder.

Conservative treatment includes transcutaneous electrical nerve stimulation (TENS), Ultrasound, LASER, Range of Motion, stretching and strengthening exercises, patient education, and home exercises. Manual therapy includes mobilization, Spencer's Muscle Energy Technique and Mobilization With Movement.

DETAILED DESCRIPTION:
The American Academy of Orthopedic Surgeons defines this condition as: "A condition of varying severity characterized by the gradual development of global limitation of active and passive shoulder motion where radiographic findings other than osteopenia are absent." Patients with frozen shoulder typically experience insidious shoulder stiffness, severe pain that usually worsens at night, and near-complete loss of passive and active external rotation of the shoulder.

Although spencer's Muscle Energy Technique is a very effective technique, still it was rarely used. It is a standardized series of steps of shoulder treatments with broad application in diagnosis, treatment, and prognosis developed by Spencer in 1961 and is a well-known osteopathic manipulative technique that focuses on mobilization of the glenohumeral and scapulothoracic joints. It is an articulatory technique in which passive, smooth, rhythmic motion of the shoulder joint is done by the therapist to stretch contracted muscles, ligaments, and capsule. Most of the force is applied at the end range of motion. This technique increases pain-free Range of Motion by stretching the tissues, enhancing lymphatic flow, and stimulating increased joint circulation.

On the other hand, "post-facilitation stretch (PFS)" is a muscle energy technique developed by Dr.Vladimir Janda to lengthen chronically shortened muscles that involves a maximal contraction of the muscle at mid-range with a rapid movement to maximal length followed by a 20-second static stretch. This technique is more aggressive than Post Isometric Relaxation and based on the concept of autogenic inhibition

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary unilateral adhesive capsulitis
* Stage II and III adhesive capsulitis
* Patients with limited active and passive Range of Motion of the affected shoulder (globally loss of at least 50% compared to non-involved shoulder in one or more directions)
* Patients with controlled diabetes

Exclusion Criteria:

* Patients with a positive history of trauma, fracture, or surgery of the cervical spine
* Corticosteroid injection in the affected shoulder in the preceding 4 weeks.
* Malignancy/Avascular Necrosis of shoulder
* Post-traumatic shoulder stiffness
* Thoracic outlet syndrome/neurological disorder
* Patients with cervical radiculopathy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
(Numeric Pain Rating Scale) | four weeks
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = the most intense pain imaginable
Goniometer | four weeks
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position. To measure the range of motion, doctors, osteopaths, physical therapists, or other health professionals most commonly use a goniometer, which is an instrument that measures angle motion at a joint
SPADI (Shoulder Pain and Disability Index) | four weeks
  The shoulder pain and disability index (SPADI) is also a reliable and valid clinimetric (Cronbach-α>0.90), self-administered questionnaire used by orthopedics and physical therapists for proper assessment of shoulder related pain and disabilities in terms of functional outcomes in patients suffering from different types of the shoulder-related pathologies. It consists of 13 items with two domains; a subscale (5-item) that measures pain, and another subscale (8-item) that assesses disability. Each subscale is added and transformed into a score that ranges from 0 (less shoulder disability) to 100 (more shoulder dysfunction).

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No